CLINICAL TRIAL: NCT05616195
Title: Application of 3D Printed Bone Prosthesis in Limb Salvage Surgery for Bone Tumors: a Single-center, Real-world Prospective Observational Study
Brief Title: Application of 3D Printed Prosthesis in Limb Salvage Surgery for Bone Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, associate chief physician, Henan Cancer Hospital
Other Study IDs: ZZUSC-18
Record Dates: First submitted 2022-10-31; First posted 2022-11-15 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-08

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3D printed bone prosthesis replacement surgery: Patients undergoing 3D-printed bone prosthesis replacement surgery
  Interventions: Other: 3D printed bone prosthesis replacement surgery

INTERVENTIONS:
Other: 3D printed bone prosthesis replacement surgery — To report the postoperative complications and limb function of patients who underwent 3D-printed bone prosthesis replacement in Henan Cancer Hospital.

SUMMARY:
To report the patients who underwent 3D-printed bone prosthesis replacement in Henan Cancer Hospital in the next 10 years, and collect the postoperative complications and limb function of these patients.

DETAILED DESCRIPTION:
To report the patients who underwent 3D-printed bone prosthesis replacement in Henan Cancer Hospital in the next 10 years. The basic data, treatment methods, postoperative complications and limb function of these patients were collected.

ELIGIBILITY:
Inclusion Criteria:

Men and women of all ages are welcome.

Pathologically confirmed in our hospital as a subtype of malignant tumor.

He received 3D printed bone prosthesis replacement in our hospital.

Exclusion Criteria:

Not applicable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing 3D-printed bone prosthesis replacement surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-28 (Estimated); Primary Completion 2032-11-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
complications | From surgery to 24 months after surgery
  Complications were collected from patients who underwent 3D-printed bone prosthesis replacement surgery.
Limb function | Patients were enrolled until 24 months after surgery
  Limb function was assessed using the Musculoskeletal Oncology Society (MSTS) scoring scale for seven items, namely movement, pain, stability, deformity, strength, functional activity, and emotional receptiveness. The highest possible score is 35, with 5 points allocated to each project.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No